CLINICAL TRIAL: NCT05299177
Title: Feasibility of Automated Insulin Delivery With an Interoperable Algorithm Using an Alternative Insulin Pump
Acronym: BELIEVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device not available
Sponsor: Imperial College London (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20HH5892
Record Dates: First submitted 2022-02-17; First posted 2022-03-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Automated Insulin Delivery (Experimental): The components of the automated insulin delivery system are the Dexcom G6 continuous glucose monitor (CGM), the InControl algorithm and an insulin pump (Ypsomed Ypsopump). The Dexcom G6 continuous glucose monitoring device is an approved device and is licensed to be used to inform insulin dosing decisions without confirmation. The algorithm (inControl 1.0) is approved when used embedded in the Tandem X2 insulin pump. We are using the algorithm for its intended purpose but are implementing it in a smartphone app to be installed in a compatible smartphone (Android). We are additionally assessing incremental benefit with the next software version of the algorithm. This will be the first time this updated software has been assessed in people with type 1 diabetes. The compatible insulin pump is a continuous subcutaneous insulin infusion device and is being used in line with its intended purpose, according to the manufacturer's instructions (YpsoMed Ypsopump).
  Interventions: Device: InControl

INTERVENTIONS:
Device: InControl — Automated insulin delivery system comprising continuous glucose sensor (Dexcom G6), controller (InControl embedded in smartphone app) and insulin pump (YpsoMed Ypsopump)

SUMMARY:
This clinical study assesses the feasibility of implementing the inControl automated insulin delivery algorithm with Dexcom continuous glucose monitoring and a compatible insulin pump in adults with type 1 diabetes. It additionally provides pilot efficacy outcomes for interoperable automated insulin delivery.

DETAILED DESCRIPTION:
Self-management of type 1 diabetes is challenging, efforts to optimise time spent in the target range can result in hypo- and hyperglycaemia. Structured education, glucose monitoring and advances in insulin delivery can increase time in range and reduce exposure to extremes of glucose and recent data confirm that automated insulin delivery can enable further increases in time spent in the target range of 3.9 to 10mmol/L (70 - 180mg/dL).

The inControl algorithm, developed by TypeZero technologies is embedded in the Tandem X2 insulin pump and operates with the Dexcom G6 continuous glucose sensor and transmitter in a CE-marked and commercially available system (known as Control-IQ). This system optimises time in range compared with sensor-augmented pump therapy, and the improvement was maintained when participants were further randomised to predictive low glucose suspend or automated insulin delivery. The United States Food and Drug Administration has defined interoperable standards for automated insulin delivery systems, including the iCGM designation for continuous glucose sensors, the interoperable automated glycaemic controller designation, and alternate controller enabled insulin pumps. However, while standards have been defined, to date, interoperability of automated insulin delivery components has not been demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Type 1 diabetes confirmed on the basis of clinical features
* Type 1 diabetes for greater than 1 year
* On an intensified insulin regimen with multiple dose injection or insulin pump for > 3 months
* HbA1c >7.5% (58mmol/mol) (or %TIR 3.9-10mmol/L <52% for participants already using a continuous glucose sensor)

Exclusion Criteria:

* Total daily insulin dose greater than 100 units
* Weight greater than 140kg
* Pregnant or planning pregnancy
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Use of any automated insulin delivery system
* Unable to participate due to other factors, as assessed by the Chief Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
% time spent in target glucose range measured by continuous glucose monitoring (3.9-10mmol/L, 70-180mg/dL) | Extracted from the final 28 days of the intervention period
  Consensus measure of time in range

SECONDARY OUTCOMES:
% time spent in hypoglycaemia (<3.0mmol/L, 54mg/dL) | Extracted from the final 28 days of the intervention period
  Consensus measure of time in range
% time spent in hypoglycaemia (<3.9mmol/L, 70mg/dL) | Extracted from the final 28 days of the intervention period
  Consensus measure of time in range
% time in euglycaemia (3.9-7.8mmol/L, 70-140mg/dL) | Extracted from the final 28 days of the intervention period
  Consensus measure of time in range
% time spent in hyperglycaemia (>10mmol/L, 180mg/dL) | Extracted from the final 28 days of the intervention period
  Consensus measure of time in range
Number hypoglycaemic excursions (sensor glucose <3.0mmol/l for >= 20min) | Over 12 week intervention period
  Consensus measure of exposure to hypoglycaemia
Nocturnal Severe hypoglycaemia (defined as requiring third party assistance) | Over 12 week intervention period
  Consensus measure of exposure to hypoglycaemia
Severe hypoglycaemia (defined as requiring third party assistance) | Over 12 week intervention period
  Consensus measure of exposure to hypoglycaemia
Glucose variability assessed by %Coefficient of Variation (%CV) | Extracted from the final 28 days of the intervention period
  Consensus measure of glucose variability
Glucose variability assessed by Mean Absolute Glucose (MAG) | Extracted from the final 28 days of the intervention period
  Consensus measure of glucose variability
Glucose variability assessed by Low Blood Glucose Index (LBGI) | Extracted from the final 28 days of the intervention period
  Consensus measure of glucose variability
HbA1c | At end of 12 week intervention period
  Laboratory HbA1c assessment
Time spent in automated insulin delivery mode | Over 12 week intervention period
  % of total time that automated insulin delivery is active
Treatment satisfaction (DTSQ, AP acceptability) | At end of 12 week intervention period
  Validated patient reported outcome
Gold score | At end of 12 week intervention period
  Validated patient reported outcome of hypoglycaemia awareness (1-7, with greater value indicating loss of awareness)
Diabetes distress (DDS-17) | At end of 12 week intervention period
  Validated patient reported outcome, Diabetes Distress Score 17 item, higher scores mean greater distress
Diabetes distress (PAID) | At end of 12 week intervention period
  Validated patient reported outcome, Problem Areas In Diabetes 20 item
Change in total daily insulin dose (units) | At end of 12 week intervention period
  Total insulin delivered by system per day
Change in weight (kg) | At end of 12 week intervention period
  Weight in kg

OTHER OUTCOMES:
Direct Resource Utilisation Costs | Over 12 week intervention period
  Health economic modelling exploratory outcome
Indirect Costs | Over 12 week intervention period
  Health economic modelling exploratory outcome
Productivity lost | Over 12 week intervention period
  Health economic modelling exploratory outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No